CLINICAL TRIAL: NCT02802423
Title: A Multi-Center, Randomized, Double Blind, Placebo-Controlled, Phase IIA Study to Evaluate the Safety and Efficacy of BLEX 404 Oral Liquid With Adjuvant Chemotherapy in Patients With Triple Negative Breast Cancer (TNBC) After Surgery
Brief Title: Phase I/II, Evaluate the Safety and Efficacy of BLEX 404 With Docetaxel in Patients With Advanced/Metastatic Triple Negative Breast Cancer.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI-1401-2-01
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; Breast cancer; Triple negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BLEX 404 Oral Liquid (Experimental): During Phase I study (dose escalation), a standard 3+3 design will be followed, and the dose range is 3 to 10 mg/kg BID. The recommended dose level (RDL) for the Phase II study is defined as the dose level with 0 to 1 DLT observed during cycle I of Docetaxel monotherapy among 6 patients in the Phase I study.
  Interventions: Drug: BLEX 404 Oral Liquid

INTERVENTIONS:
Drug: BLEX 404 Oral Liquid — BLEX 404 Oral Liquid is administered twice daily during the Docetaxel monotherapy period. The dose of Docetaxel is 75 mg/m2 IV, 21 days a cycle.

SUMMARY:
The primary purpose of this study is to determine the safety and recommended dose level (RDL) of BLEX 404 Oral Liquid combined with Docetaxel monotherapy in a 21-day schedule. The secondary purpose is to assess the efficacy and safety of BLEX 404 Oral Liquid combined with Docetaxel monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 20 - 70 years old at the time of signing the ICF.
2. Patients with histologically or pathologically diagnosed with advanced/metastatic triple negative (ER-, PR-, and HER2-negative) breast cancer.

   1. ER =< 10% by immunohistochemistry (IHC) tumor staining;
   2. PR =< 10% by IHC tumor staining;
   3. HER2-negative defined as one of the following: 0 or 1+ by IHC, or 2+ by IHC and fluorescence in situ hybridization (FISH)-negative (ratio < 2.0).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Adequate hematologic function defined as: absolute neutrophil count (ANC) greater than or equal to 2,000/μL; platelets count greater than or equal to 100,000/μL; hemoglobin must be greater than or equal to 10 g/dL (can be corrected by growth factor or transfusion).
5. Adequate hepatic function defined as: serum bilirubin less than or equal to 1.5-fold upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) less than or equal to 3-fold ULN.
6. Adequate renal function with: serum creatinine less than or equal to 1.3 mg/dL or calculated creatinine clearance greater than or equal to 60 mL/minute according to the Cockcroft and Gault formula.
7. Women must be either of non-child bearing potential, or women with child-bearing potential agree to use effective a highly contraceptive method or a contraceptive implant, exception of hormonal contraception (estrogen/progesterone), from time of Screening Visit until 30 days after study drug discontinuation.
8. Planning to receive Docetaxel monotherapy.
9. Willing and able to comply with all aspects of the treatment protocol.
10. Provide written informed consent.

Exclusion Criteria:

1. Patient with brain metastasis.
2. Patient with autoimmune disease that requires systemic steroids or immunosuppression agents.
3. Current enrollment in another clinical study or used any investigational drug or device within the past 28 days preceding informed consent.
4. Patients with following treatment prior to Docetaxel monotherapy: chemotherapy, immunotherapy, or biologic systemic anticancer therapy within 21 days of study entry (42 days for mitomycin and nitrosoureas); prior taxanes; radiation therapy within 28 days (3 months for bone marrow exposure 20%); hormonal therapy within 4 weeks.
5. Known history of human immunodeficiency virus (HIV) infection.
6. Existing anticancer treatment-related toxicities of Grades greater than or equal to 2 (except for alopecia and neuropathy) according to Common Terminology Criteria for Adverse Events (CTCAE v4.03).
7. Patients with Grade > 2 neuropathy.
8. Patient has an active infection requiring systemic therapy.
9. History of concomitant medical conditions or infectious diseases that, in the opinion of the investigator, would compromise the subject's ability to safely complete the study.
10. Clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolonged QT/QTc ([QT interval/corrected QT interval].
11. Ascertained hypersensitivity to any component of investigational product used in the study.
12. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily BLEX 404 Oral Liquid treatment.
13. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation, psychiatric disorder, with any other serious diseases/medical history.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicity (DLT) observation | 3 weeks (1 cycle)
  Presence or absence of dose-limiting toxicity (DLT) related to BLEX 404 Oral Liquid for each patient during first cycle of Docetaxel monotherapy to determine the recommended dose level (RDL).
Phase II: Overall response rate (PR + CR) | 12 weeks (4 cycles)
  Overall response rate (PR + CR) after 4 cycles of combination use in BLEX 404 + Docetaxel monotherapy.

SECONDARY OUTCOMES:
Phase II: Overall response rate (PR + CR)(at least 1 cycle) | at least 3 weeks (1 cycle)
  Overall response rate (PR + CR) after at least 1 cycle of combination use in BLEX 404 + Docetaxel monotherapy.
Phase II: Incidence of grade 3/4 hematological toxicity | 3 weeks (1 cycle)
  Rate of grade 3/4 hematological toxicity of each cycle.
Quality of Life by EORTC QLQ-C30 | 3 weeks (1 cycle)
  Examination of quality of life by EORTC QLQ-C30 questionnaire of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Richard King, Ph.D., Study Director — American BriVision Corporation